CLINICAL TRIAL: NCT04531761
Title: Evaluating the Efficacy of the Parent Support Program
Acronym: PSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Em Matsuno, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2019-116
Record Dates: First submitted 2020-08-17; First posted 2020-08-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Prejudice; Gender Identity; Knowledge, Attitudes, Practice
Keywords: transgender; trans youth; parental acceptance; parental support; LGBTQ
MeSH Terms: conditions — Prejudice; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Access to Parent Support Program (Experimental)
  Interventions: Behavioral: Parent Support Program
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Parent Support Program — The parent support program includes three modules aimed at increasing knowledge, positive attitudes, and supportive behaviors towards trans youth. Each online module includes several activities including writing prompts, videos, interactive quizzes, and other educational activities.
  Arms: Immediate Access to Parent Support Program

SUMMARY:
The objective of the study is to evaluate the efficacy of an online intervention (the Parents Support Program) aimed at increasing supportive behaviors among parents of transgender youth. The intervention consists of three modules that include a variety engaging activities such as social perspective taking exercises, writing prompts, videos of parents, youth, and experts, and psycho-educational materials. The study uses an experimental design with a waitlist control. Both the experimental and control groups will complete a pre-test, one month follow up, and two month follow up survey. Targeted outcomes include knowledge about gender diversity, attitudes about trans youth, and supportive parenting behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must live in the United States.
* Must be comfortable communicating in English.
* Must be a parent of a trans child between the ages of 10 - 24.

Exclusion Criteria:

* Participants who participated in pilot study or focus groups related to this project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Trans-supportive behaviors scale | One month
  This 20 item questionnaire measures the frequency of supportive behaviors enacted in the past month. Response options ranged from 1 (never) to 5 (frequently) based on item anchors from the Ryan et al. (2010) measure on family acceptance. The original 25-item scale was reduced to 20 items based on achieving adequate internal consistency reliability in a previous study with parents of trans youth (Matsuno & Israel, in preparation). An example item is: "I told my child I respect and support them." The measure showed adequate internal consistency reliability in the pilot study of the Parent Support Program (α = .8).

SECONDARY OUTCOMES:
Attitudes Toward Trans Youth Scale (ATTYS - Birnkrant, 2018) | One month
  Two subscales of the original scale were used consisting of 27 items- Genderism, and Fabricated Identity. The scale had strong reliablity α = .98 and demonstrated convergent and discriminant validity.
Objective knowledge about gender diversity | One month
  The author created a 18-item measure designed to test knowledge about constructs of gender and experiences of transgender people. The items are based on the program content and through best practices for creating multiple choice questions.
Subjective knowledge about gender diversity | One month
  Participants perceptions of their own level knowledge regarding gender diversity will be measured using a 100-point Likert scale from 1 - not at all knowledgeable to 100- extremely knowledgeable. Participants will be asked to rate their perceived knowledge in the following areas: gender terminology, etiology, medical intervention, and impact of parental acceptance.
Self-compassion | One month
  Self-compassion was measured by adapting the self-kindness subscale of the Self-Compassion Scale - Short Form (SCS-SF) (Raes, Pommier, Neff, & Van Gucht, 2011). The subscale demonstrated adequate reliability in a previous sample (α = .78) (Raes et al., 2011). The five items were adapted by adding "as a parent of a trans/non-binary child" at the end of each item to measure self-compassion related to parenting a trans child. Items were rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). The measure showed strong internal consistency reliability in the pilot study of the Parent Support Program (α = .94).

CONTACTS AND LOCATIONS:
Overall Officials: Em Matsuno, PhD, Principal Investigator — Palo Alto University
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.